CLINICAL TRIAL: NCT02981342
Title: An Adaptive, Open-Label, Randomized Phase 2 Study of Abemaciclib as a Monotherapy and in Combination With Other Agents Versus Choice of Standard of Care (Gemcitabine or Capecitabine) in Patients With Previously Treated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of Abemaciclib (LY2835219) Alone or in Combination With Other Agents in Participants With Previously Treated Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16342; I3Y-MC-JPCJ (Other: Eli Lilly and Company); 2016-002218-36 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-08-18

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — abemaciclib; LY3023414; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abemaciclib (Experimental): Abemaciclib given orally.
  Interventions: Drug: Abemaciclib
- Abemaciclib + LY3023414 (Experimental): Abemaciclib given orally and LY3023414 given orally.
  Interventions: Drug: Abemaciclib; Drug: LY3023414
- Standard of Care (Gemcitabine or Capecitabine) (Experimental): Gemcitabine given intravenously (IV) OR capecitabine given orally.
  Interventions: Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib; Abemaciclib + LY3023414
Drug: LY3023414 — Administered orally
  Arms: Abemaciclib + LY3023414
Drug: Gemcitabine — Administered IV
  Other Names: LY188011
  Arms: Standard of Care (Gemcitabine or Capecitabine)
Drug: Capecitabine — Administered orally
  Arms: Standard of Care (Gemcitabine or Capecitabine)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of abemaciclib alone and in combination with other drugs versus standard of care in participants with previously treated metastatic pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of ductal adenocarcinoma of the pancreas.
* Metastatic disease with documented disease progression following previous treatment with at least one, but no more than 2 prior therapies, with one of the prior therapies having been either gemcitabine-based or fluoropyrimidine-based therapy. Neoadjuvant and/or adjuvant therapies for localized resectable or unresectable PDAC each count as a line of therapy if multiagent chemotherapy regimens were administered (and neoadjuvant regimen was different than adjuvant regimen) and if the participant progressed with metastatic disease while taking or within 6 months of completion of (neo)adjuvant therapy.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant for whom treatment with monotherapy chemotherapy such as gemcitabine or capecitabine is a reasonable choice.
* Discontinued all prior treatment for cancer at least 14 days prior to initial dose of study treatment.
* Adequate organ function.

  * allow alanine aminotransferase (ALT) or aspartate aminotransferase (AST) up to 5x upper limit of normal (ULN) if liver metastases.
  * allow bilirubin up to 2.5 times ULN if elevation is not associated with other signs of liver toxicity or can be explained by mechanical obstruction - requires clinical research physician approval.

Exclusion Criteria:

* Have a personal history of any of the following conditions: syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Exception: Participants with controlled atrial fibrillation for >30 days prior to study treatment initiation are eligible.
* Have insulin-dependent diabetes mellitus. Participants with type 2 diabetes mellitus are eligible if adequate control of blood glucose level is obtained by oral anti-diabetics as documented by hemoglobin A1c (HbA1c) <7%.
* Have symptomatic central nervous system metastasis. Screening of asymptomatic participants is not required for enrollment.
* Have had major surgery within 7 days prior to initiation of study drug to allow for postoperative healing of the surgical wound and site(s).
* Have previously received treatment with any cyclin-dependent kinase (CDK) 4 and 6 inhibitor or phosphatidylinositol 3-kinase (PI3K) and/or mammalian target of rapamycin (mTOR) inhibitor or have a known hypersensitivity to any component of the investigational products in this study.
* Have a known hypersensitivity to investigator's choice of standard of care (gemcitabine or capecitabine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (30):
- United States (10):
  - Yale University School of Medicine, New Haven, Connecticut
  - Illinois CancerCare, Peoria, Illinois
  - Research Medical Center, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Olympia, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Blacktown
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edegem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Wilrijk
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramat Gan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L'Hospitalet de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - Fundacion Jimenez Diaz, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
  More information provided by Eli Lilly and Company
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chiorean EG, Picozzi V, Li CP, Peeters M, Maurel J, Singh J, Golan T, Blanc JF, Chapman SC, Hussain AM, Johnston EL, Hochster HS. Efficacy and safety of abemaciclib alone and with PI3K/mTOR inhibitor LY3023414 or galunisertib versus chemotherapy in previously treated metastatic pancreatic adenocarcinoma: A randomized controlled trial. Cancer Med. 2023 Oct;12(20):20353-20364. doi: 10.1002/cam4.6621. Epub 2023 Oct 16. PMID 37840530
- See also: A Study of Abemaciclib (LY2835219) Alone or in Combination with Other Agents in Participants with Previously Treated Pancreatic Ductal Adenocarcinoma — https://www.lillytrialguide.com/en-US/studies/pancreatic-ductal-adenocarcinoma/JPCJ#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was planned for stage 1 & stage 2. No participants were enrolled to stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled to stage 1.
  Completed participants are those who has CR, PR, SD, or PD and is off treatment.
Pre-assignment Details: Per protocol, no efficacy analysis was planned for safety lead in. Purpose of safety lead in was only safety evaluation. All efficacy was done on randomized pts.
Groups:
- 150mg Abemaciclib + 150mg Galunisertib (Safety Lead-in): Participants received oral dose of 150mg Abemaciclib twice daily for 28 day cycles along with oral dose of 150 mg Galunisertib twice daily for 14 days of 28 days cycle.
- 200mg Abemaciclib: Participants received oral dose of 200mg Abemaciclib twice daily (BID) for 28 day cycles.
- 150mg Abemaciclib + 150mg LY3023414: Participants received oral dose of 150mg Abemaciclib along with 150mg LY3023414 twice daily for 28 day cycles.
- Gemcitabine or Capecitabine: Participants received either 1000 milligram per square meter (mg/m^2) of Gemcitabine by intravenous infusion on days 1, 8, 15 and 22 of 28 day cycle or 1250 mg/m^2 oral dose of Capecitabine twice daily for 14 days of 21 day cycle.
Period: Overall Study
Arm/Group | 150mg Abemaciclib + 150mg Galunisertib (Safety Lead-in) | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Started | 7 | 33 | 33 | 33
Received at Least One Dose of Study Drug | 7 | 32 | 33 | 26
Completed | 7 | 22 | 20 | 19
Not Completed | 0 | 11 | 13 | 14
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 0 | 9 | 9 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1
Not completed — Study closed by sponsor | 0 | 0 | 1 | 1
Not completed — Randomized, Never Treated | 0 | 1 | 0 | 7
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150mg Abemaciclib + 150mg Galunisertib (Safety Lead-in) | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine | Total
Number analyzed (Participants) | 7 | 33 | 33 | 33 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants who received at least one dose of study drug.
  years
    number analyzed (Participants) | 7 | 32 | 33 | 26 | 98
    (all) | 65.29 (6.99) | 61.09 (7.83) | 62.52 (8.97) | 66.85 (7.61) | 63.40 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 18 | 16 | 19 | 57
  Male | 3 | 15 | 17 | 14 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 3 | 9
  Not Hispanic or Latino | 7 | 30 | 28 | 24 | 89
  Unknown or Not Reported | 0 | 1 | 1 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 7 | 5 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 3 | 4
  White | 7 | 26 | 26 | 25 | 84
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 8 | 6 | 5 | 19
  United States | 7 | 8 | 10 | 8 | 33
  Taiwan | 0 | 7 | 4 | 3 | 14
  United Kingdom | 0 | 1 | 0 | 0 | 1
  Israel | 0 | 2 | 4 | 5 | 11
  Australia | 0 | 1 | 1 | 3 | 5
  France | 0 | 1 | 1 | 6 | 8
  Spain | 0 | 5 | 7 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Disease control rate (DCR) is the percentage of participants with a best overall response of CR, PR or SD as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anticancer Therapy (Up to 6 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 33 | 33 | 33
percentage of Participants | 15.2 [2.9 to 27.4] | 12.1 [1.0 to 23.3] | 36.4 [20 to 52.8]
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.0495, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.0230, Cochran-Mantel-Haenszel

2. Primary Outcome: Stage 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until first observation of objective progressive disease as defined by RECIST v1.1 or death from any cause, whichever comes first. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a patient does not have a complete baseline disease assessment, then the PFS time will be censored at the randomization date, regardless of whether or not objectively determined disease progression or death has been observed for the patient; otherwise, if a patient is not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time will be censored at the last complete objective progression-free disease assessment date.
Time Frame: Baseline to Measured Progressive Disease or Death Due to Any Cause (Up to 6 Months)
Population: All randomized participants. Censored participants: Abemaciclib 200 mg: 3, Abemaciclib 150mg + LY3023414 150mg: 8, Gemcitabine & Capecitabine: 18; No participants were enrolled in stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled in stage 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 33 | 33 | 33
Months | 1.68 [1.35 to 1.84] | 1.81 [1.28 to 1.91] | 3.25 [1.05 to 5.65]
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.0085, Log Rank
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.0123, Log Rank

3. Secondary Outcome: Stage 1: Objective Response Rate (ORR): Percentage of Participants With a Best Overall Response (BOR) of CR or PR
Description: Objective response rate (ORR) is the percentage of participants with a BOR of CR or PR as defined by RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline to Measured Progressive Disease or Start of New Anti-Cancer Therapy (Up to 6 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 33 | 33 | 33
percentage of Participants | 3 [0 to 8.9] | 0 [NA to NA] — Data did not allow it to be estimable. | 3 [0 to 8.9]
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.3017, Cochran-Mantel-Haenszel

4. Secondary Outcome: Stage 1: Pharmacokinetics (PK): Mean Steady State Exposure of Abemaciclib and Its Metabolites (LSN2839567 (M2), LSN3106726 (M20))
Description: Mean steady state exposure was reported as measured by maximum observed plasma concentration (Cmax).
Time Frame: Cycle(C)1 Day(D)14: 0 hour(h),0.5h,1h,2h,4h,6h,8h post dose
Population: All randomized participants who received at least one dose of Abemaciclib along with Galunisertib and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Millilitre (ng/mL)
Groups:
- 150mg Abemaciclib + 150mg Galunisertib: Participants received oral dose of 150mg Abemaciclib twice daily for 28 day cycles along with oral dose of 150 mg Galunisertib twice daily for 14 days of 28 days cycle.
Arm/Group | 150mg Abemaciclib + 150mg Galunisertib
Number analyzed (Participants) | 4
Nanogram per Millilitre (ng/mL)
  Abemaciclib | 356 (137)
  LSN2839567 (M2) | 85.1 (66)
  LSN3106726 (M20) | 153 (58)

5. Secondary Outcome: Stage 1: PK: Area Under the Curve (AUC) (AUC[Tau]) of LY3023414
Time Frame: Cycle 1 Day 1 through Cycle 4 Day 1 (28 Day Cycles)
Population: Zero Participants Analyzed: AUC cannot be calculated due to insufficient data collected.
Arm/Group | 150mg Abemaciclib + 150mg LY3023414
Number analyzed (Participants) | 0

6. Secondary Outcome: Stage 1: PK: Maximum Concentration (Cmax) at Steady State of LY3023414
Time Frame: Cycle 1 Day 1 through Cycle 4 Day 1 (28 Day Cycles)
Population: Zero Participants Analyzed: Cmax cannot be calculated due to insufficient data collected.
Arm/Group | 150mg Abemaciclib + 150mg LY3023414
Number analyzed (Participants) | 0

7. Secondary Outcome: Stage 2: Disease Control Rate (DCR): Percentage of Participants With a Best Overall Response of CR, PR, and SD
Time Frame: Baseline to Measured Progressive Disease or Start of New Anticancer Therapy (Up to 6 Months)
Population: Data not reported, no patients were enrolled to stage 2.
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Stage 2: Clinical Benefit Rate (CBR): Percentage of Participants With Best Overall Response of CR, PR, or SD With Duration of SD for at Least 6 Months
Description: Clinical benefit rate (CBR) is the percentage of participants with a BOR of CR or PR, or SD ≥6 months. CR is defined as the disappearance of all target and non-target lesions & no appearance of new lesions. PR is defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
  No participants were enrolled to stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled to stage 1.
Time Frame: Baseline to Disease Progression or Start of New Anticancer Therapy (Up to 6 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants | 3 [0 to 8.9] | 0 [0 to 0] | 3 [0 to 8.9]
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.3017, Cochran-Mantel-Haenszel

9. Secondary Outcome: Stage 2: Duration of Response (DoR)
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Up to 6 Months)
Population: The population for analyzing DoR is the number of participants with response of CR or PR. There was only one participant in 200 mg Abemaciclib arm and one participant in Gemcitabine/Capecitabine arm. Due to small number of participants, the data is not analyzable using the planned time to event analysis.
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Stage 2: Overall Survival (OS)
Description: OS duration is measured from the date of randomization to the date of death from any cause. for participants who is not known to have died as of the data-inclusion cutoff date, OS was censored at the last known alive date.
  No participants were enrolled to stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled to stage 1.
Time Frame: Baseline to Death from Any Cause (Up to 10 Months)
Population: All randomized participants. Censored participants: Abemaciclib 200mg: 11, Abemaciclib 150mg + LY3023414 150mg: 12, Gemcitabine + Capecitabine: 21;
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 33 | 33 | 33
Months | 2.71 [1.97 to 5.36] | 3.29 [1.97 to 5.03] | NA [2.53 to NA] — Data did not allow it to be estimable.
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.1938, Log Rank; Hazard Ratio (HR) = 1.600, 95% CI 2-sided [0.782 to 3.272]
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.2477, Log Rank; Hazard Ratio (HR) = 1.533, 95% CI 2-sided [0.746 to 3.150]

11. Secondary Outcome: Stage 2: Change From Baseline in Carbohydrate Antigen 19.9 (CA 19-9) Level
Description: No participants were enrolled to stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled to stage 1.
Time Frame: Baseline, 6 Months
Population: All randomized participants with baseline and post baseline CA 19-9 measurement.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 24 | 21 | 20
U/mL | 4281.53 (8177.89) | 3225.29 (5730.25) | -501.17 (7198.70)

12. Secondary Outcome: Stage 2: Change From Baseline in Pain and Symptom Burden Assessment on the Modified Brief Pain Inventory-Short Form (mBPI-sf)
Description: mBPI-sf is an 11-item instrument used as a multiple-item measure of cancer pain intensity. In addition to pain intensity (4 items), the mBPI-sf is designed for participants to record the presence of pain in general, pain relief, and pain interference with function (general activity, mood, ability to walk, ability to perform normal work, relations with others, sleep, and enjoyment of life). Responses for the mBPI-sf items are captured through the use of 11-point numeric rating scales anchored at 0 (no pain or does not interfere) and ranged through 10 (pain as bad as you can imagine or completely interferes). The mBPI-sf recall period is 24 hours, and typical completion time for this instrument is less than 5 minutes.
  No participants were enrolled to stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled to stage 1.
Time Frame: Baseline, 6 Months
Population: All randomized participants with baseline & post baseline value for the mBPI-sf specified item.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 19 | 14 | 13
score on a scale
  Pain at its Worst in Last 24 hours | 0.63 (0.47) | -0.33 (0.55) | -0.02 (0.57)
  Pain at its Least in Last 24 hours | 0.86 (0.42) | 0.18 (0.49) | 0.39 (0.51)
  Pain on the Average: number analyzed (Participants) | 18 | 14 | 13
  Pain on the Average | 0.62 (0.45) | -0.03 (0.51) | -0.07 (0.53)
  Pain Right Now | 0.38 (0.34) | 0.34 (0.59) | -0.38 (0.61)
  Pain Interfered General Activity | 0.64 (0.47) | 0.07 (0.55) | 0.22 (0.57)
  Pain Interfered with Mood | 0.54 (0.41) | 0.28 (0.48) | 0.60 (0.50)
  Pain Interfered Walking Ability | 0.05 (0.55) | 0.83 (0.64) | 0.19 (0.67)
  Pain Interfered with Normal Work | 1.07 (0.51) | 0.66 (0.59) | 0.19 (0.61)
  Pain Interfered with Relations | 0.39 (0.52) | 0.67 (0.61) | 0.26 (0.63)
  Pain Interfered with Sleep | 0.19 (0.53) | 0.34 (0.61) | -0.56 (0.65)
  Pain Interfered Enjoyment of Life | 0.69 (0.62) | 0.39 (0.72) | -0.13 (0.75)
  BPI Mean Pain Interference Score | 0.55 (0.44) | 0.50 (0.51) | 0.05 (0.54)
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain at its Worst in Last 24 Hours; Test type: Superiority; p = 0.383, Mixed Models Analysis; LSMean Difference = 0.65, 95% CI 2-sided [-0.84 to 2.13], Standard Error of Mean 0.74
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain at its Worst in Last 24 Hours; Test type: Superiority; p = 0.692, Mixed Models Analysis; LSMean Difference = -0.31, 95% CI 2-sided [-1.91 to 1.28], Standard Error of Mean 0.79
Statistical Analysis 3: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain at its Least in Last 24 Hours; Test type: Superiority; p = 0.469, Mixed Models Analysis; LSMean Difference = 0.48, 95% CI 2-sided [-0.85 to 1.80], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain at its Least in Last 24 Hours; Test type: Superiority; p = 0.776, Mixed Models Analysis; LSMean Difference = -0.20, 95% CI 2-sided [-1.62 to 1.22], Standard Error of Mean 0.70
Statistical Analysis 5: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain on the Average; Test type: Superiority; p = 0.328, Mixed Models Analysis; LSMean Difference = 0.69, 95% CI 2-sided [-0.72 to 2.11], Standard Error of Mean 0.70
Statistical Analysis 6: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain on the Average; Test type: Superiority; p = 0.954, Mixed Models Analysis; LSMean Difference = 0.04, 95% CI 2-sided [-1.45 to 1.54], Standard Error of Mean 0.74
Statistical Analysis 7: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Right Now; Test type: Superiority; p = 0.350, Mixed Models Analysis; LSMean Difference = 0.75, 95% CI 2-sided [-0.85 to 2.36], Standard Error of Mean 0.80
Statistical Analysis 8: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain right now; Test type: Superiority; p = 0.405, Mixed Models Analysis; LSMean Difference = 0.72, 95% CI 2-sided [-1.01 to 2.44], Standard Error of Mean 0.85
Statistical Analysis 9: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered General Activity; Test type: Superiority; p = 0.565, Mixed Models Analysis; LSMean Difference = 0.43, 95% CI 2-sided [-1.06 to 1.91], Standard Error of Mean 0.73
Statistical Analysis 10: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain Interfered General Activity; Test type: Superiority; p = 0.848, Mixed Models Analysis; LSMean Difference = -0.15, 95% CI 2-sided [-1.74 to 1.43], Standard Error of Mean 0.79
Statistical Analysis 11: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered with Mood; Test type: Superiority; p = 0.928, Mixed Models Analysis; LSMean Difference = -0.06, 95% CI 2-sided [-1.37 to 1.25], Standard Error of Mean 0.65
Statistical Analysis 12: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain Interfered with Mood; Test type: Superiority; p = 0.650, Mixed Models Analysis; LSMean Difference = -0.32, 95% CI 2-sided [-1.71 to 1.08], Standard Error of Mean 0.69
Statistical Analysis 13: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered Walking Ability; Test type: Superiority; p = 0.865, Mixed Models Analysis; LSMean Difference = -0.15, 95% CI 2-sided [-1.89 to 1.60], Standard Error of Mean 0.86
Statistical Analysis 14: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain Interfered Walking Ability; Test type: Superiority; p = 0.497, Mixed Models Analysis; LSMean Difference = 0.63, 95% CI 2-sided [-1.23 to 2.50], Standard Error of Mean 0.92
Statistical Analysis 15: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered with Normal Work; Test type: Superiority; p = 0.272, Mixed Models Analysis; LSMean Difference = 0.89, 95% CI 2-sided [-0.72 to 2.50], Standard Error of Mean 0.80
Statistical Analysis 16: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain Interfered with Normal Work; Test type: Superiority; p = 0.583, Mixed Models Analysis; LSMean Difference = 0.47, 95% CI 2-sided [-1.25 to 2.19], Standard Error of Mean 0.85
Statistical Analysis 17: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered with Relations; Test type: Superiority; p = 0.876, Mixed Models Analysis; LSMean Difference = 0.13, 95% CI 2-sided [-1.53 to 1.79], Standard Error of Mean 0.82
Statistical Analysis 18: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered with relations; Test type: Superiority; p = 0.644, Mixed Models Analysis; LSMean Difference = 0.41, 95% CI 2-sided [-1.37 to 2.19], Standard Error of Mean 0.88
Statistical Analysis 19: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered with Sleep; Test type: Superiority; p = 0.384, Mixed Models Analysis; LSMean Difference = 0.75, 95% CI 2-sided [-0.97 to 2.48], Standard Error of Mean 0.85
Statistical Analysis 20: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Test type: Superiority; p = 0.318, Mixed Models Analysis; LSMean Difference = 0.90, 95% CI 2-sided [-0.90 to 2.71], Standard Error of Mean 0.89
Statistical Analysis 21: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Pain Interfered Enjoyment of Life; Test type: Superiority; p = 0.407, Mixed Models Analysis; LSMean Difference = 0.81, 95% CI 2-sided [-1.15 to 2.78], Standard Error of Mean 0.97
Statistical Analysis 22: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Pain Interfered Enjoyment of Life; Test type: Superiority; p = 0.620, Mixed Models Analysis; LSMean Difference = 0.52, 95% CI 2-sided [-1.58 to 2.62], Standard Error of Mean 1.04
Statistical Analysis 23: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; BPI-Mean Interference Score; Test type: Superiority; p = 0.475, Mixed Models Analysis; LSMean Difference = 0.50, 95% CI 2-sided [-0.90 to 1.91], Standard Error of Mean 0.70
Statistical Analysis 24: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; BPI-Mean Interference Score; Test type: Superiority; p = 0.540, Mixed Models Analysis; LSMean Difference = 0.46, 95% CI 2-sided [-1.04 to 1.96], Standard Error of Mean 0.74

13. Secondary Outcome: Stage 2: Change From Baseline in Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 self-reported general cancer instrument consists of 30 items covered by 1 of 3 dimensions:
  1. Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  2. Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much)
  3. Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function/QOL or higher levels of symptom burden.
  No participants were enrolled to stage 2; however, results for stage 2 outcomes are reported from the data collected for participants enrolled to stage 1.
Time Frame: Baseline, 6 Months
Population: All randomized participants with baseline & post baseline value for the EORTC QLQ-C30 specified item.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
Number analyzed (Participants) | 19 | 14 | 14
units on a scale
  Global Health Status: number analyzed (Participants) | 19 | 14 | 13
  Global Health Status | -6.21 (3.87) | -4.82 (4.50) | -2.40 (4.64)
  Functional Scales: Physical Functioning | -14.44 (4.40) | -11.65 (5.12) | -5.42 (5.12)
  Functional Scales: Role Functioning | -17.09 (6.17) | -18.05 (7.32) | -17.10 (7.36)
  Functional Scales: Emotional Functioning: number analyzed (Participants) | 19 | 14 | 13
  Functional Scales: Emotional Functioning | -4.89 (4.49) | -0.63 (5.22) | 2.06 (5.41)
  Functional Scales: Cognitive Functioning: number analyzed (Participants) | 19 | 14 | 13
  Functional Scales: Cognitive Functioning | -10.43 (4.10) | -8.39 (4.77) | -5.18 (4.95)
  Functional Scale: Social Functioning: number analyzed (Participants) | 19 | 14 | 13
  Functional Scale: Social Functioning | -21.12 (4.90) | -17.09 (5.72) | -2.00 (5.95)
  Symptom Scales: Fatigue | 14.13 (4.92) | 14.90 (5.73) | 5.64 (5.71)
  Symptom Scales: Nausea and Vomiting | 7.98 (5.57) | 9.42 (6.47) | 11.88 (6.50)
  Symptom Scales: Pain | 9.79 (5.63) | 2.68 (6.61) | 5.43 (6.62)
  Symptom Scale: Dysopnea | 0.35 (5.48) | 11.19 (6.38) | -4.51 (6.36)
  Symptom Scale: Insomnia | -5.19 (5.17) | 1.83 (6.01) | -6.71 (6.05)
  Symptom Scale: Appetite Loss: number analyzed (Participants) | 19 | 14 | 12
  Symptom Scale: Appetite Loss | 12.54 (5.79) | 15.32 (6.77) | 9.51 (7.30)
  Symptom Scale: Constipation: number analyzed (Participants) | 19 | 14 | 13
  Symptom Scale: Constipation | 2.96 (5.95) | -6.51 (6.96) | 12.93 (7.15)
  Symptom Scale: Diarrhoea: number analyzed (Participants) | 19 | 14 | 13
  Symptom Scale: Diarrhoea | 15.71 (6.76) | 26.28 (7.83) | 20.51 (7.98)
  Symptom Scale: Financial difficulties: number analyzed (Participants) | 19 | 14 | 13
  Symptom Scale: Financial difficulties | 3.96 (4.82) | 2.45 (5.68) | -3.30 (5.87)
Statistical Analysis 1: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Global health status; Test type: Superiority; p = 0.818, Mixed Models Analysis; LSMean Difference = -1.39, 95% CI 2-sided [-13.46 to 10.68], Standard Error of Mean 5.98
Statistical Analysis 2: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Global health status; Test type: Superiority; p = 0.533, Mixed Models Analysis; LSMean Difference = -3.80, 95% CI 2-sided [-16.03 to 8.42], Standard Error of Mean 6.06
Statistical Analysis 3: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Functional Scales: Physical functioning; Test type: Superiority; p = 0.681, Mixed Models Analysis; LSMean Difference = -2.79, 95% CI 2-sided [-16.40 to 10.82], Standard Error of Mean 6.75
Statistical Analysis 4: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Functional Scales: Physical functioning; Test type: Superiority; p = 0.189, Mixed Models Analysis; LSMean Difference = -9.02, 95% CI 2-sided [-22.63 to 4.59], Standard Error of Mean 6.75
Statistical Analysis 5: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Functional Scales: Role functioning; Test type: Superiority; p = 0.921, Mixed Models Analysis; LSMean Difference = 0.96, 95% CI 2-sided [-18.29 to 20.21], Standard Error of Mean 9.54
Statistical Analysis 6: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Functional Scales: Role functioning; Test type: Superiority; p = 0.999, Mixed Models Analysis; LSMean Difference = 0.01, 95% CI 2-sided [-19.40 to 19.42], Standard Error of Mean 9.62
Statistical Analysis 7: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Functional Scales: Emotional functioning; Test type: Superiority; p = 0.541, Mixed Models Analysis; LSMean Difference = -4.26, 95% CI 2-sided [-18.20 to 9.68], Standard Error of Mean 6.91
Statistical Analysis 8: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Functional Scales: Emotional functioning; Test type: Superiority; p = 0.330, Mixed Models Analysis; LSMean Difference = -6.95, 95% CI 2-sided [-21.17 to 7.27], Standard Error of Mean 7.05
Statistical Analysis 9: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Functional Scales: Cognitive Functioning; Test type: Superiority; p = 0.747, Mixed Models Analysis; LSMean Difference = -2.04, 95% CI 2-sided [-14.74 to 10.66], Standard Error of Mean 6.29
Statistical Analysis 10: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Functional Scales: Cognitive functioning; Test type: Superiority; p = 0.419, Mixed Models Analysis; LSMean Difference = -5.25, 95% CI 2-sided [-18.22 to 7.73], Standard Error of Mean 6.43
Statistical Analysis 11: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Functional Scales: Social functioning; Test type: Superiority; p = 0.596, Mixed Models Analysis; LSMean Difference = -4.02, 95% CI 2-sided [-19.23 to 11.19], Standard Error of Mean 7.53
Statistical Analysis 12: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Functional Scales: Social functioning; Test type: Superiority; p = 0.017, Mixed Models Analysis; LSMean Difference = -19.12, 95% CI 2-sided [-34.68 to -3.55], Standard Error of Mean 7.71
Statistical Analysis 13: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptoms Scales: Fatigue; Test type: Superiority; p = 0.919, Mixed Models Analysis — Social Scales: Fatigue; LSMean Difference = -0.77, 95% CI 2-sided [-16.03 to 14.49], Standard Error of Mean 7.57
Statistical Analysis 14: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Fatigue; Test type: Superiority; p = 0.267, Mixed Models Analysis; LSMean Difference = 8.48, 95% CI 2-sided [-6.72 to 23.69], Standard Error of Mean 7.54
Statistical Analysis 15: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Nausea and Vomiting; Test type: Superiority; p = 0.866, Mixed Models Analysis; LSMean Difference = -1.45, 95% CI 2-sided [-18.66 to 15.77], Standard Error of Mean 8.54
Statistical Analysis 16: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Nausea and Vomiting; Test type: Superiority; p = 0.652, Mixed Models Analysis; LSMean Difference = -3.90, 95% CI 2-sided [-21.23 to 13.43], Standard Error of Mean 8.59
Statistical Analysis 17: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Pain; Test type: Superiority; p = 0.417, Mixed Models Analysis; LSMean Difference = 7.11, 95% CI 2-sided [-10.39 to 24.60], Standard Error of Mean 8.67
Statistical Analysis 18: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Pain; Test type: Superiority; p = 0.618, Mixed Models Analysis; LSMean Difference = 4.36, 95% CI 2-sided [-13.16 to 21.89], Standard Error of Mean 8.69
Statistical Analysis 19: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Dyspnoea; Test type: Superiority; p = 0.206, Mixed Models Analysis; LSMean Difference = -10.84, 95% CI 2-sided [-27.85 to 6.18], Standard Error of Mean 8.44
Statistical Analysis 20: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Dyspnoea; Test type: Superiority; p = 0.566, Mixed Models Analysis; LSMean Difference = 4.86, 95% CI 2-sided [-12.08 to 21.80], Standard Error of Mean 8.40
Statistical Analysis 21: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Insomnia; Test type: Superiority; p = 0.380, Mixed Models Analysis; LSMean Difference = -7.02, 95% CI 2-sided [-23.01 to 8.96], Standard Error of Mean 7.93
Statistical Analysis 22: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Insomnia; Test type: Superiority; p = 0.850, Mixed Models Analysis; LSMean Difference = 1.52, 95% CI 2-sided [-14.60 to 17.64], Standard Error of Mean 7.99
Statistical Analysis 23: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Appetite loss; Test type: Superiority; p = 0.756, Mixed Models Analysis; LSMean Difference = -2.79, 95% CI 2-sided [-20.78 to 15.21], Standard Error of Mean 8.91
Statistical Analysis 24: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Appetite loss; Test type: Superiority; p = 0.747, Mixed Models Analysis; LSMean Difference = 3.02, 95% CI 2-sided [-15.77 to 21.82], Standard Error of Mean 9.31
Statistical Analysis 25: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Constipation; Test type: Superiority; p = 0.311, Mixed Models Analysis; LSMean Difference = 9.47, 95% CI 2-sided [-9.16 to 28.09], Standard Error of Mean 9.23
Statistical Analysis 26: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Constipation; Test type: Superiority; p = 0.290, Mixed Models Analysis; LSMean Difference = -9.97, 95% CI 2-sided [-28.75 to 8.80], Standard Error of Mean 9.30
Statistical Analysis 27: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Diarrhoea; Test type: Superiority; p = 0.323, Mixed Models Analysis; LSMean Difference = -10.57, 95% CI 2-sided [-31.93 to 10.78], Standard Error of Mean 10.58
Statistical Analysis 28: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Diarrhoea; Test type: Superiority; p = 0.651, Mixed Models Analysis; LSMean Difference = -4.80, 95% CI 2-sided [-26.08 to 16.48], Standard Error of Mean 10.54
Statistical Analysis 29: Comparison: 200mg Abemaciclib vs Gemcitabine or Capecitabine; Symptom Scales: Financial Difficulties; Test type: Superiority; p = 0.841, Mixed Models Analysis; LSMean Difference = 1.51, 95% CI 2-sided [-13.57 to 16.59], Standard Error of Mean 7.47
Statistical Analysis 30: Comparison: 150mg Abemaciclib + 150mg LY3023414 vs Gemcitabine or Capecitabine; Symptom Scales: Financial Difficulties; Test type: Superiority; p = 0.344, Mixed Models Analysis; LSMean Difference = 7.26, 95% CI 2-sided [-8.03 to 22.54], Standard Error of Mean 7.57

14. Secondary Outcome: Stage 1: PK: Steady State Trough Pre Dose Concentration of LY3023414
Description: Mean steady state exposure was reported by trough pre-dose plasma concentrations.
Time Frame: C2D1: 0h, C3D1: 0h, C4D1: 0h
Population: All randomized participants who received at least one dose of 150mg LY3023414 and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 150mg Abemaciclib + 150mg LY3023414: Participants received oral dose of 150mg Abemaciclib twice daily along with 150mg LY3023414 twice daily for 28 day cycles.
Arm/Group | 150mg Abemaciclib + 150mg LY3023414
Number analyzed (Participants) | 9
ng/mL | 27.3 (450)

15. Secondary Outcome: Stage 1: PK: Mean Single Dose Concentration of LY3023414 at 2h Post-dose
Description: Mean single dose exposure was reported by plasma concentrations collected approximately 2 hours post-dose.
Time Frame: C1D1: 2h Post dose
Population: All randomized participants who received at least one dose of 150mg LY3023414 and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 150mg Abemaciclib + 150mg LY3023414
Number analyzed (Participants) | 28
ng/mL | 518 (67)

ADVERSE EVENTS:
Time Frame: Up to 30 weeks
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- 150mg Abemaciclib + 150mg Galunisertib (Safety Lead - In): Participants received oral dose of 150mg Abemaciclib twice daily for 28 day cycles along with oral dose of 150 mg Galunisertib twice daily for 14 days of 28 days cycle.
Arm/Group | 150mg Abemaciclib + 150mg Galunisertib (Safety Lead - In) | 200mg Abemaciclib | 150mg Abemaciclib + 150mg LY3023414 | Gemcitabine or Capecitabine
All-Cause Mortality (participants affected / at risk) | 5/7 | 22/32 | 21/33 | 12/26
Serious Adverse Events (participants affected / at risk) | 4/7 | 17/32 | 18/33 | 15/26
Other Adverse Events (participants affected / at risk) | 7/7 | 30/32 | 33/33 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150mg Abemaciclib + 150mg Galunisertib (Safety Lead - In) (N=7) | 200mg Abemaciclib (N=32) | 150mg Abemaciclib + 150mg LY3023414 (N=33) | Gemcitabine or Capecitabine (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 150mg Abemaciclib + 150mg Galunisertib (Safety Lead - In) (N=7) | 200mg Abemaciclib (N=32) | 150mg Abemaciclib + 150mg LY3023414 (N=33) | Gemcitabine or Capecitabine (N=26)
Anaemia (Blood and lymphatic system disorders) | 3 (14) | 10 (18) | 6 (7) | 11 (19)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (9) | 0 (0) | 2 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (17)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (8) | 5 (5) | 6 (8)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (2) | 5 (6) | 2 (2) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 12 (21) | 17 (19) | 8 (16)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 9 (14) | 15 (18) | 9 (10)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 12 (16) | 6 (9)
Vomiting (Gastrointestinal disorders) | 2 (3) | 10 (12) | 15 (22) | 6 (8)
Asthenia (General disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (7) | 16 (22) | 17 (25) | 11 (12)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 4 (4) | 5 (6) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (5) | 5 (6) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (8) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (6) | 0 (0) | 1 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 5 (9) | 3 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 5 (16) | 1 (1) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1) | 1 (2) | 3 (5) | 1 (3)
Blood potassium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 2 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (7) | 1 (3) | 2 (8)
Occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 10 (20) | 5 (11) | 4 (9)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3) | 4 (4) | 1 (3) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 9 (11) | 8 (9) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (5) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 3 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (4) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (3) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 3 (6) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0/3 (0) | 0/14 (0) | 1/17 (1) | 0/10 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (5) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 10 (24)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 3 (3) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was planned for stage 1 & stage 2. Stage 2 did not occur, no participants were enrolled to stage 2;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02981342/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT02981342/SAP_001.pdf